CLINICAL TRIAL: NCT05657886
Title: The Effect of Half Swaddle and Kangaroo Care Practıces Initiated in The Early Period In Preterm Infants on Breastfeeding, Mother-Infant Attachment, Maternal Sleep Quality and Postpartum Depression
Brief Title: Half Swaddle and Kangaroo Care in Preterm on Breastfeeding, Infant Attachment, Sleep Quality and Depression of Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Research Assistant, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020/P0226
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Kangaroo Care
Keywords: Breastfeeding; Mother-infant attachment; Maternal sleep quality; Postpartum depression; Half swaddle
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): The mothers in the control group were given routine care.
- Half swaddle (Experimental): HS applied to a newborn baby makes the baby feel completely safe, as if in the womb. After laying the soft fabric or baby blanket, it was placed in the supine position. Half swaddling was done so as not to restrict the baby's arm and leg movements. HS was performed 15 minutes before each sleep during the day until the 3rd month.
  Interventions: Other: Half swaddle
- Kangaroo care (Experimental): The application was applied at twice a day and for 60 min, every day for 6 months in a row. While the mothers were taken to the NICU and practiced at home prior to kangaroo care, hand hygiene and breast care were provided within the scope of infection prevention rules. During KC, the mother placed her baby between two breasts, and the baby's breast was placed on the mother's breast in an upright position. During the application of KC, a quiet, calm and suitable environment was created so that comfort of the baby and mother would not be disturbed. The mother and baby are covered with a blanket. The ambient temperature was 26 centigrade degrees during the kangaroo care. In the continuation of the KB application, the mother was asked to breastfeed her baby. In order to prevent the risk of aspiration of the baby after breastfeeding, the baby was placed in the left lateral position so that the mother and the baby could lie down together.
  Interventions: Other: Kangaroo care
- Half swaddle+Kangaroo care (Experimental): HS applied to a newborn baby makes the baby feel completely safe, as if in the womb. After laying the soft fabric or baby blanket, it was placed in the supine position. Half swaddling was done so as not to restrict the baby's arm and leg movements. HS was performed 15 minutes before each sleep during the day until the 3rd month.The application was applied at twice a day and for 60 min, every day for 6 months in a row. During KC, the mother placed her baby between two breasts, and the baby's breast was placed on the mother's breast in an upright position. During the application of KC, a quiet, calm and suitable environment was created so that comfort of the baby and mother would not be disturbed. The mother and baby are covered with a blanket. In the continuation of the KB application, the mother was asked to breastfeed her baby.
  Interventions: Other: Half swaddle; Other: Kangaroo care

INTERVENTIONS:
Other: Half swaddle — Half swaddle: HS applied to a newborn baby makes the baby feel completely safe, as if in the womb. After laying the soft fabric or baby blanket, it was placed in the supine position. Half swaddling was done so as not to restrict the baby's arm and leg movements. HS was performed 15 minutes before each sleep during the day until the 3rd month.
  Arms: Half swaddle; Half swaddle+Kangaroo care
Other: Kangaroo care — The application was applied twice a day and for 60 minutes every day for 6 months in a row. During KC, the mother placed her baby between two breasts, and the baby's breast was placed on the mother's breast in an upright position. During the application of KC, a quiet, calm, and the suitable environment was created so that comfort of the baby and mother would not be disturbed. The mother and baby are covered with a blanket. The ambient temperature was 26 centigrade degrees during the kangaroo care. In the continuation of the KB application, the mother was asked to breastfeed her baby. In order to prevent the risk of aspiration of the baby after breastfeeding, the baby was placed in the left lateral position so that the mother and the baby could lie down together. The researcher observed the application steps of the mother's KC, and the deficiencies, if any, were corrected by discussing with the mother during/after the application.
  Arms: Half swaddle+Kangaroo care; Kangaroo care

SUMMARY:
Aim: The aim of this study is to investigate the effect of half swaddle and kangaroo care practices initiated in the early period in preterm infants on breastfeeding, mother-infant attachment, maternal sleep quality and postpartum depression.

Design: The prospective, randomized controlled study

DETAILED DESCRIPTION:
The prospective, randomized controlled study was conducted on 160 mothers with premature babies whose age were between 18 and 49 randomly divided into four groups as 40 case group, 40 half swaddle group, 40 kangaroo care group, 40 half swaddle and kangaroo care group at the neonatal intensive care service and birth service of Trakya University Health Research and Application Center between September 2020 and March 2022.

In order to determine the number of samples, in order to test the difference in the effect size of 0.3326851 calculated between the groups based on the 1-month difference in the EPDS scores in the study of Herizchi et al. (2017), with 5% margin of error and 95% power, a total of n=40 from each group was used. It was calculated that the mothers who gave =160 preterm births should be included in the study.

N=160 samples of preterm infants were randomized with the help of ASS 11 (NCSS, LLC. Kaysville, Utah. www.ncss.com) computer program, HS group (n=40), KC group (n=40), HS+KC group. (n=40) and control (n=40) groups.

Data were collected using Survey Form, Edinburgh Postpartum Depression Scale (EPDS), Pittsburgh Sleep Quality Index (PSQI), Mother-to-Infant Bonding Scale (MIBS), Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), Latch Breastfeeding Diagnosis Measurement Form, Perception of Insufficient Milk Questionnaire (PIMQ). Data were evaluated using descriptive analyses, Mann Whitney U, Kruskal Wallis Test, Friedman S Test, Spearmen Correlation, multiple linear regression analysis.

Research data It was collected using the Survey Form, Edinburgh Postpartum Depression Scale (EPDS), Pittsburgh Sleep Quality Index (PSQI), Mother-to-Infant Bonding Scale (MIBS), Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), Latch Breastfeeding Diagnosis Measurement Form, Perception of Insufficient Milk Questionnaire (PIMQ).

Survey form; It which was prepared by the researchers by reviewing the literature consists of 5 main sections and a total of 82 questions, including the personal characteristics of the mother who gave birth preterm, the characteristics of the birth and the baby, the characteristics of sleep, the characteristics of the baby's sleep pattern, and the characteristics of the baby's growth and development.

Edinburgh Postnatal Depression Scale (EPDS): The scale was developed by Cox and Holden (1987). Adapted to Turkish by Engindeniz, Küey, and Kültür (1996). It is used to determine the risk for depression in the postnatal period and to measure the level and change of violence. It is a self-assessment scale. It is applied to postpartum women. It contains a total of 10 questions and measures depression. It provides a four-point Likert type measurement. The directive is at the beginning of the scale and subjects are asked to mark the substance most relevant to their situation when filling in the subjects. The total score of the scale is obtained by adding these item scores. As a result of the cut-off point scale study conducted in Turkey and it has ben calculated as 12/13

Pittsburgh Sleep Quality Index (PSQI): PSQI is a self-reported screening and assessment questionnaire that details information on the type and severity of sleep quality and disorders within the last month. It was developed by Buysse et al. (20), and its validity and reliability study in Turkish was performed by Agargün et al. (21). PUKI evaluates sleep quality in the last month. 18 items and 7 components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, daytime dysfunction) are included in the scoring. Each item is evaluated over 0-3 points and the sum of 7 component points gives the total PUKI score. The total score ranges from 0 to 21, with higher scores indicating worsening sleep quality. A total PUKI score of ≤5 is considered "good sleep", and >5 is considered "bad sleep".

Mother-to-Infant Bonding Scale (MIBS): MIBS was developed by Taylor et al.12. The MIBS is a measurement tool that can be applied easily and quickly by the puerperal from the first day of the postpartum period and that allows the mother to express her feelings for her baby. This scale shows the relationship between the bond between mother and infant and the mother's mood during the early postpartum period. The MIBS is a four-point Likert-type scale consisting of eight items. Answers are scored between 0-3, the lowest score that can be obtained from the scale is 0 and the highest score is 24. High scores indicate a problem with mother-infant bonding. A Turkish validity and reliability study of the scale was conducted by Karakulak and Alparslan.

Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF): The BSES-SF was developed by Dennis (1999). Later, the short form of the scale was developed by Dennis (2003) by reducing it. The BSES-SF is a 14-item instrument developed to measure breastfeeding confidence. All the items are preceded by the statement "I can always" and are anchored by a five-point Likert-type scale, with 1 = not at all confident and 5 = always confident. All the items are presented positively and the scores are summed up to produce a final score ranging from 14 to 70, with the higher scores indicating better BSE. Turkish validity and reliability of the scale were done by Tokat and Okumuş (2013).

Latch Breastfeeding Diagnosis Measurement Form: It is a measurement tool developed by Jensen et al. (1994). The Turkish validity of the Latch Breastfeeding Diagnosis Measurement Form was performed by Yenal and Okumus (2003). The Latch Breastfeeding Diagnosis Measurement Form consists of the combination of the first letters of the English equivalent of the five evaluation criteria and is listed as follows: L (Latch on breast), A (Audible swallowing), T (Type of nipple), C (Comfort breast/nipple), H (Hold / Help). Each item in the scale is evaluated between 0-2 points. The lowest 0 and the highest 10 points are obtained from the scale. Total high score indicates the baby's sucking success.

Perception of Insufficient Milk Questionnaire (PIMQ): Designed based on the conceptual model of McCarter-Spaulding and Kearney (2001), clinical experience, and literature, this six-question questionnaire was designed to measure the perception of insufficient milk in breastfeeding mothers. Turkish validity and reliability study was done by Gökçeoğlu. The first question is a ''yes'' or ''no'' question about whether them other perceives her milk as sufficient and other questions assess whether the mother perceives her milk as insufficient. Mothers rated these questions between 0 and 10, with ''0" meaning that her milk is perceived as completely insufficient, and ''10" meaning that her milk is perceived as completely sufficient. The lowest and highest scores possible on the scale are 0 and 50, respectively. The value of the total score indicates how high the score is and whether the perception of the amount of milk is sufficient.

Data collection The mean scores of BSES-SF, IMPS, LATCH, MIAS, PSQI and EPDS at the beginning, 1st, 2nd, 3rd and 6th months of the half swaddling and kangaroo care group

Intervention. Half swaddle: HS applied to a newborn baby makes the baby feel completely safe, as if in the womb. After laying the soft fabric or baby blanket, it was placed in the supine position. Half swaddling was done so as not to restrict the baby's arm and leg movements. HS was performed 15 minutes before each sleep during the day until the 3rd month.

Kangaroo care: The application was applied at twice a day and for 60 min, every day for 6 months in a row. While the mothers were taken to the NICU and practiced at home prior to kangaroo care, hand hygiene and breast care were provided within the scope of infection prevention rules. During KC, the mother placed her baby between two breasts, and the baby's breast was placed on the mother's breast in an upright position. During the application of KC, a quiet, calm and suitable environment was created so that comfort of the baby and mother would not be disturbed. The mother and baby are covered with a blanket. The ambient temperature was 26 centigrade degrees during the kangaroo care. In the continuation of the KB application, the mother was asked to breastfeed her baby. In order to prevent the risk of aspiration of the baby after breastfeeding, the baby was placed in the left lateral position so that the mother and the baby could lie down together. The application steps of the mother's KC were observed by the researcher and the deficiencies, if any, were corrected by discussing with the mother during / after the application.

Control group: The mothers in the control group were given routine care.

ELIGIBILITY:
Inclusion Criteria:

For the mother;

* Volunteer to participate in the research,
* Over 18 years old,
* Had a preterm birth (single birth less than 38 weeks),
* After an uncomplicated pregnancy process, the delivery was completed by normal vaginal or cesarean delivery method,
* Prepregnancy BMI <35,
* Stable vital signs, For baby;
* Birth weight below 2500 g,
* Stable vital signs,
* APGAR score of 7 and above,
* Hospitalized for a minimum of 5 days,
* Babies who are 2 weeks or more postpartum.

Exclusion Criteria:

For the mother;

* Over 49 years old,
* Full-term birth (38-42 weeks single birth),
* Using cigarettes, alcohol and stimulants,
* Pre-pregnancy BMI>35,
* Working night shift,
* Having received infertility treatment,
* Having a chronic disease (such as hypertension, diabetes mellitus),
* Experiencing severe depression, anxiety and stress,
* Having any organic or non-organic disease that may cause cognitive impairment (such as Delirium, Dementia, Intellectual Retardation),
* Mothers with serious maternal complications,

For baby;

* Birth weight of 2500 g and above,
* APGAR score below 7,
* Having serious neonatal complications,
* Congenital malformation,
* Hospitalized for a maximum of 5 days,
* Babies under 2 weeks postpartum.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2020-07-05 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
breastfeeding evaluated using the Breastfeeding Self-Efficacy Scale-Short Form | change from before implamentation patent and 1st, 2nd, 3rd, and 6th months of practice.
  ): The BSES-SF was developed by Dennis (1999). Later, the short form of the scale was developed by Dennis (2003) by reducing it. The BSES-SF is a 14-item instrument developed to measure breastfeeding confidence. All the items are preceded by the statement "I can always" and are anchored by a five-point Likert-type scale, with 1 = not at all confident and 5 = always confident. All the items are presented positively and the scores are summed up to produce a final score ranging from 14 to 70, with the higher scores indicating better BSE. Turkish validity and reliability of the scale were done by Tokat and Okumuş (2013).
breastfeeding evaluated using the Latch Breastfeeding Diagnosis Measurement Form | change from before implamentation patent and 1st, 2nd, 3rd, and 6th months of practice.
  It is a measurement tool developed by Jensen et al. (1994). The Turkish validity of the Latch Breastfeeding Diagnosis Measurement Form was performed by Yenal and Okumus (2003). The Latch Breastfeeding Diagnosis Measurement Form consists of the combination of the first letters of the English equivalent of the five evaluation criteria and is listed as follows: L (Latch on breast), A (Audible swallowing), T (Type of nipple), C (Comfort breast/nipple), H (Hold / Help). Each item in the scale is evaluated between 0-2 points. The lowest 0 and the highest 10 points are obtained from the scale. Total high score indicates the baby's sucking success.
breastfeeding evaluated using the Perception of Insufficient Milk Questionnaire (PIMQ) | change from before implamentation patent and 1st, 2nd, 3rd, and 6th months of practice.
  Designed based on the conceptual model of McCarter-Spaulding and Kearney (2001), clinical experience, and literature, this six-question questionnaire was designed to measure the perception of insufficient milk in breastfeeding mothers. Turkish validity and reliability study was done by Gökçeoğlu. The first question is a ''yes'' or ''no'' question about whether them other perceives her milk as sufficient and other questions assess whether the mother perceives her milk as insufficient. Mothers rated these questions between 0 and 10, with ''0" meaning that her milk is perceived as completely insufficient, and ''10" meaning that her milk is perceived as completely sufficient. The lowest and highest scores possible on the scale are 0 and 50, respectively. The value of the total score indicates how high the score is and whether the perception of the amount of milk is sufficient.
mother infant attachment evaluated using the Mother-to-Infant Bonding Scale (MIBS) | change from before implamentation patent and 1st, 2nd, 3rd, and 6th months of practice.
  MIBS was developed by Taylor et al.12. The MIBS is a measurement tool that can be applied easily and quickly by the puerperal from the first day of the postpartum period and that allows the mother to express her feelings for her baby. This scale shows the relationship between the bond between mother and infant and the mother's mood during the early postpartum period. The MIBS is a four-point Likert-type scale consisting of eight items. Answers are scored between 0-3, the lowest score that can be obtained from the scale is 0 and the highest score is 24. High scores indicate a problem with mother-infant bonding. A Turkish validity and reliability study of the scale was conducted by Karakulak and Alparslan.
mother sleep quality evaluated using the Pittsburgh Sleep Quality Index (PSQI) | change from before implamentation patent and 1st, 2nd, 3rd, and 6th months of practice.
  PSQI is a self-reported screening and assessment questionnaire that details information on the type and severity of sleep quality and disorders within the last month. It was developed by Buysse et al. (20), and its validity and reliability study in Turkish was performed by Agargün et al. (21). PUKI evaluates sleep quality in the last month. 18 items and 7 components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, daytime dysfunction) are included in the scoring. Each item is evaluated over 0-3 points and the sum of 7 component points gives the total PUKI score. The total score ranges from 0 to 21, with higher scores indicating worsening sleep quality. A total PUKI score of ≤5 is considered "good sleep", and >5 is considered "bad sleep".
postpartum depression evaluated using the Edinburgh Postnatal Depression Scale (EPDS) | change from before implamentation patent and 1st, 2nd, 3rd, and 6th months of practice.
  The scale was developed by Cox and Holden (1987). Adapted to Turkish by Engindeniz, Küey, and Kültür (1996). It is used to determine the risk for depression in the postnatal period and to measure the level and change of violence. It is a self-assessment scale. It is applied to postpartum women. It contains a total of 10 questions and measures depression. It provides a four-point Likert type measurement. The directive is at the beginning of the scale and subjects are asked to mark the substance most relevant to their situation when filling in the subjects. The total score of the scale is obtained by adding these item scores. As a result of the cut-off point scale study conducted in Turkey and it has ben calculated as 12/13.

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey, Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided